CLINICAL TRIAL: NCT05526664
Title: Omics Gaucher Study: Multiomic Approach To Describe The Gaucher Disease Treatment Dynamics In Comparison To Untreated Healthy Volunteers
Brief Title: Omics Gaucher Study: Multiomic Approach
Acronym: OmicsGaucher
Status: Active, not recruiting | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: OG 01-2022
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-09

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Gaucher Type 1: * The participant was diagnosed with Gaucher type 1 disease
  * Adults only
  Interventions: Other: Genetic testing and Omics analysis
- Gaucher Type 3: * The participant was diagnosed with Gaucher type 3 disease
  * Adults only
  Interventions: Other: Genetic testing and Omics analysis
- Healthy Volunteer: * Healthy participants
  * Adults only
  Interventions: Other: Genetic testing and Omics analysis

INTERVENTIONS:
Other: Genetic testing and Omics analysis — Blood sample for genetic analysis and for Omics analysis as metabolomics and transcriptomics

SUMMARY:
The study aims to investigate the transcriptomic and metabolomic changes in blood, plasma and isolated monocytes from Gaucher patients and healthy controls.

DETAILED DESCRIPTION:
Gaucher disease is one of the most common lysosomal storage disorders (LSD) and is an autosomal recessive inherited disorder, primed by mutation in the GBA1 gene which leads to a deficiency in β-glucocerebrosidase (GCase) activity and accumulation of its substrate glucosylceramide (GluCer)/-sphingosine (GluSph). The macrophages are the main cell type exhibiting a Gaucher disease phenotype. The large accumulation of GluCer and to a lesser extent that of GluSph lead to dysfunction in organs such as spleen, liver, bone marrow, and lungs.

However, a validated, reproducible, and broadly applicable tool to classify Gaucher Disease at any stage of the disease is still missing.

The development of new technologies, such as genomic analysis by next generation sequencing (NGS) and other "omics technologies," has advanced the molecular understanding and diagnosis of Rare Diseases

The current study will analyze the transcriptional and metabolomic profiles in blood, plasma and isolated monocytes from Gaucher patients and healthy controls with the aim to compare these profiles and to define how much a patient profile differs from a healthy one.

ELIGIBILITY:
Inclusion Criteria:

Gaucher Type 1 participants:

* Informed consent
* The participant is older than 18 years old
* The participant was diagnosed with Gaucher Type 1 disease

Gaucher Type 3 participants:

* Informed consent
* The participant is older than 18 years old
* The participant was diagnosed with Gaucher type 3 disease

Healthy participants:

* Informed consent
* The participant is older than 18 years old
* Healthy participants

Exclusion Criteria:

Gaucher Type I participants:

* The participant had any other clinically significant disease
* The participant had a recent (within 14 days) acute infection and/or vaccination

Gaucher Type 3 participants:

* Diagnosis of a significant CNS disease or cardiovascular disease other than Gaucher type 3
* The participant had a recent (within 14 days) acute infection and/or vaccination

Healthy participants:

* The participant had a recent (within 14 days) acute infection and/or vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gaucher participants diagnosed with Type 1 and Type 3. Healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
OMICS DATA | 12 months
  investigate the transcriptomic and metabolomic changes in blood, plasma and isolated monocytes from Gaucher patients and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, MD, Principal Investigator — CENTOGENE GmbH
Locations (1):
- UKE, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No